CLINICAL TRIAL: NCT04457336
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Efficacy and Safety of SPR001 (Tildacerfont) in Adult Subjects With Classic Congenital Adrenal Hyperplasia
Brief Title: A Ph2b to Evaluate Clinical Efficacy and Safety of Tildacerfont in Adult CAH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study SPR001-203 did not meet its primary and secondary endpoints therefore Spruce Biosciences has decided to terminate the study
Sponsor: Spruce Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPR001-203; CAHmelia 203 (Other: Spruce Biosciences)
Record Dates: First submitted 2020-06-25; First posted 2020-07-07 (Actual); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: CAH; Adrenal Disorder; Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Adrenal Gland Diseases

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1:1:1 manner to one of three doses of Tildacerfont or Placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Tildacerfont Group 1 (Experimental): Tildacerfont administered daily via oral tablet for 12 weeks at dose level 1
  Interventions: Drug: Tildacerfont/Placebo
- Tildacerfont Group 2 (Experimental): Tildacerfont administered daily via oral tablet for 12 weeks at dose level 2
  Interventions: Drug: Tildacerfont/Placebo
- Tildacerfont Group 3 (Experimental): Tildacerfont administered daily via oral tablet for 70 weeks at dose level 3
  Interventions: Drug: Tildacerfont/Placebo
- Placebo (Placebo Comparator): Placebo administered daily via oral tablet for 12 weeks.
  Interventions: Drug: Tildacerfont/Placebo

INTERVENTIONS:
Drug: Tildacerfont/Placebo — Tablet, administered daily
  Other Names: SPR001

SUMMARY:
An investigation of the efficacy and safety of up to 70 weeks of treatment with Tildacerfont in subjects with classic CAH who have elevated biomarkers at baseline on their current GC regimen. Optional open label treatment extension period up to 240 weeks with 200mg Tildacerfont QD.

DETAILED DESCRIPTION:
This is a study that will test the efficacy and safety of Tildacerfont. The first 12-weeks will be a double-blind, placebo controlled, dose ranging study. The following 58-weeks will assess the long term safety of Tildacerfont. Optional open label treatment extension period up to 240 weeks with 200mg Tildacerfont QD.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥18 years old at screening
2. Has a known childhood diagnosis of classic CAH due to 21-hydroxylase deficiency based on genetic mutation in CYP21A2 and/or documented (at any time) elevated 17-OHP and currently treated with HC, HC acetate, prednisone, prednisolone, methylprednisolone (or a combination of the aforementioned GCs)
3. Has been on a stable, supraphysiologic dose of GC replacement (defined as ≥15 mg/day and ≤60 mg/day in HCe) for ≥1 month before screening
4. Has A4 >ULN at both screening and Week 4 (measured before any AM GC dose) if daily GC dose <30 mg OR has A4 >2.5x ULN at both screening and Week 4 (measured before any AM GC dose)
5. For subjects with the salt-wasting form of CAH, subject has been on a stable dose of mineralocorticoid replacement for ≥1 month before screening
6. Agrees to follow contraception guidelines. Male subjects must also agree to refrain from donating sperm throughout the treatment period and for 90 days after the last dose of study drug.
7. Is able to understand all study procedures and risks involved and provides written informed consent indicating willingness to comply with all aspects of the protocol.

Exclusion Criteria:

1. Has a known or suspected diagnosis of any other known form of classic CAH (not due to 21 hydroxylase deficiency)
2. Has a history that includes bilateral adrenalectomy or hypopituitarism
3. Has a history of allergy or hypersensitivity to tildacerfont, any of its excipients, or any other CRF1 receptor antagonist
4. Current treatment with dexamethasone as GC therapy for CAH

   a. Prior treatment with dexamethasone is allowed as long as the transition to an alternative GC regimen (eg, HC, prednisone, or prednisolone) has resulted in a stable dose of GC replacement for ≥1 month before screening.
5. Is not adherent to GC or study drug dosing regimen during the Run-in Period (defined as taking <80% of expected doses based on drug accountability)
6. Shows clinical signs or symptoms of adrenal insufficiency
7. Has had a clinically significant unstable medical condition, medically significant illness, or chronic disease occurring within 30 days of screening, including but not limited to:

   1. An ongoing malignancy or <3 years of remission history from any malignancy, other than successfully treated localized skin cancer
   2. eGFR of <45 mL/min/1.73 m2
   3. Current or history of liver disease (with the exception of Gilbert's syndrome).
   4. History of alcohol or substance abuse within the last year, or any significant history of alcohol or substance abuse that would likely prevent the subject from reliably participating in the study, based on the opinion of the Investigator
   5. Active hepatitis B, hepatitis C, or HIV at screening
   6. Subjects who plan to undergo bariatric surgery during the study are excluded.
   7. Any other condition that would impact subject safety or confound interpretation of study results
8. Psychiatric conditions, including but not limited to bipolar disorder, schizophrenia, or schizoaffective disorders that are not effectively controlled on medication and may have an adverse impact on study compliance. Symptoms including hallucinations, delusions, and psychosis are exclusionary. Additionally:

   1. Increased risk of suicide based on the Investigator's judgment or the results of the C-SSRS conducted at screening and Week 6 (eg, C-SSRS Type 3, 4, or 5 ideation within the past 6 months or any suicidal behavior within the past 12 months)
   2. HADS score >12 for either depression or anxiety at screening or Week 6
9. Has clinically significant abnormal ECG or clinical laboratory results. Abnormal results that must be reviewed and discussed with the Medical Monitor to determine eligibility for this study include but are not limited to:

   1. Any clinically meaningful abnormal ECG results, including QTcF >450 ms for male participants or >470 ms for female participants
   2. ALT >2x ULN
   3. Total bilirubin >1.5x ULN
   4. Total bile acids >5x ULN
10. Routinely works overnight shifts
11. Subjects with travel plans/work schedules that result in significant and frequent changes in time zones (>2 hours) will require Medical Monitor approval for enrollment.
12. Females who are pregnant or nursing
13. Use of any other investigational drug from 30 days or 5 half-lives (whichever is longer) before screening to the end of the study
14. Use of the following drugs from 30 days or 5 half-lives (whichever is longer) before Day 1 to the end of the study:

    1. Rosiglitazone, aromatase inhibitors, testosterone, growth hormones, or any other medication or supplement that could impact subject safety or confound interpretation of study results
    2. The following drugs:

    i. Moderate to strong inhibitors and/or inducers of CYP3A4 ii. Sensitive substrates or narrow-therapeutic-range substrates of CYP3A4 (except hormonal contraception containing ≤35 μg ethinyl estradiol) iii. Sensitive substrates or narrow-therapeutic-range substrates of BCRP (except those that can be administered QD in the morning, separated by approximately 10 hours from evening administration of study drug)
15. Donation or receipt of blood from 90 days before Screening to the end of the study; donation or receipt of platelets, white blood cells, or plasma from 30 days before Screening to the end of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyriakie Sarafoglou, M.D, Principal Investigator — Dept. of Pediatrics, Divisions of Endocrinology and Genetics & Metabolism, Univ. of Minnesota
Locations (64):
- United States (27):
  - Spruce Study Site, Birmingham, Alabama
  - Spruce Study Site, Los Angeles, California
  - Spruce Clinical Site, Orange, California
  - Spruce Study Site, Sacramento, California
  - Spruce Study Site, Englewood, Colorado
  - Spruce Clinical Site, Tampa, Florida
  - Spruce Study Site, West Palm Beach, Florida
  - Spruce Study Site, Chicago, Illinois
  - Spruce Clinical Site, Indianapolis, Indiana
  - Spruce Study Site, Baltimore, Maryland
  - Spruce Clinical Site, Minneapolis, Minnesota
  - Spruce Study Site, Rochester, Minnesota
  - Spruce Clinical Site, Las Vegas, Nevada
  - Spruce Study Site, Hickory, North Carolina
  - Spruce Study Site, Canton, Ohio
  - Spruce Study Site, Cincinnati, Ohio
  - Spruce Study Site, Cleveland, Ohio
  - Spruce Study Site, Columbus, Ohio
  - Spruce Clinical Site, Bend, Oregon
  - Spruce Study Site, Philadelphia, Pennsylvania
  - Spruce Study Site, Providence, Rhode Island
  - Spruce Study Site, Columbia, South Carolina
  - Spruce Clinical Site, Memphis, Tennessee
  - Spruce Study Site, Austin, Texas
  - Spruce Study Site, Dallas, Texas
  - Spruce Clinical Site, Edinburg, Texas
  - Spruce Clinical Site, Fort Worth, Texas
- Australia (4):
  - Spruce Study Site, Nedlands, Western Australia
  - Spruce study site, Brisbane
  - Spruce Study Site, Elizabeth Vale
  - Spruce Study Site, Melbourne
- Brazil (2):
  - Spruce Study Site, Brasília
  - Spruce Study Site, São Paulo
- Canada (4):
  - Spruce Study Site, St. John's, Newfoundland and Labrador
  - Spruce Study Site, London, Ontario
  - Spruce Study Site, Ottawa
  - Spruce Study Site, Sherbrooke
- Denmark (2):
  - Spruce Study Site, Aarhus
  - Spruce Study Site, Copenhagen
- Estonia (2):
  - Spruce Study Site, Tallinn
  - Spruce Study Site, Tartu
- Spruce Study Site, Munich, Germany
- Spruce Study Site, Dublin, Ireland
- Italy (4):
  - Spruce Study Site, Milan
  - Spruce Study Site, Napoli
  - Spruce Study Site, Rome
  - Spruce Study Site, Torino
- Spruce Study Site, Riga, Latvia
- Spruce Study Site, Kaunas, Lithuania
- Spruce Study Site, Nijmegen, Netherlands
- Poland (2):
  - Spruce Study Site, Krakow
  - Spruce Study Site, Warsaw
- Spruce Study Site, Bucharest, Romania
- Spruce Study Site, Seoul, South Korea
- Spain (4):
  - Spruce Study Site, Barcelona
  - Spruce Study Site, Madrid
  - Spruce Study Site, Seville
  - Spruce Study Site, Tarragona
- Sweden (2):
  - Spruce Study Site, Falun
  - Spruce Study Site, Stockholm
- Switzerland (2):
  - Spruce Study Site, Sankt Gallen
  - Spruce Study Site, Zurich
- Spruce Study Site, Istanbul, Turkey (Türkiye)
- Spruce Study Site, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 96 participants participated in Part A , 86 of those participants continued into Part B, and 57 of these participants then entered Part C
Pre-assignment Details: 96 informed consents were signed when participants enrolled in the Placebo or Part A of the study. The ICF included language for all Parts of the study.
Groups:
- Period 1: Placebo: Placebo
- Period 2: Part A 50 mg; Period 3: Part B 50 mg: Tildacerfont 50 mg
- Period 2: Part A 100 mg; Period 3: Part B 100 mg: Tildacerfont 100 mg
- Period 2: Part A 200 mg; Period 3: Part B 200 mg: Tildacerfont 200 mg
- Period 4: Part C: Tildacerfont tablet administered daily via oral tablet for 46 weeks at 200 mg
Period: Period 1: Placebo
Arm/Group | Period 1: Placebo | Period 2: Part A 50 mg | Period 2: Part A 100 mg | Period 2: Part A 200 mg | Period 3: Part B 50 mg | Period 3: Part B 100 mg | Period 3: Part B 200 mg | Period 4: Part C
Started | 24 | 0 (Tildacerfont treatment only) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 24 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2: Part A
Arm/Group | Period 1: Placebo | Period 2: Part A 50 mg | Period 2: Part A 100 mg | Period 2: Part A 200 mg | Period 3: Part B 50 mg | Period 3: Part B 100 mg | Period 3: Part B 200 mg | Period 4: Part C
Started | 0 | 24 | 24 | 24 | 0 | 0 | 0 | 0
Completed | 0 | 20 | 21 | 21 | 0 | 0 | 0 | 0
Not Completed | 0 | 4 | 3 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Study Terminated | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Period 3: Part B
Arm/Group | Period 1: Placebo | Period 2: Part A 50 mg | Period 2: Part A 100 mg | Period 2: Part A 200 mg | Period 3: Part B 50 mg | Period 3: Part B 100 mg | Period 3: Part B 200 mg | Period 4: Part C
Started | 0 | 0 | 0 | 0 | 1 | 44 | 41 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 33 | 26 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 11 | 15 | 0
Not completed — Study Terminated | 0 | 0 | 0 | 0 | 1 | 10 | 13 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Period: Period 4: Part C
Arm/Group | Period 1: Placebo | Period 2: Part A 50 mg | Period 2: Part A 100 mg | Period 2: Part A 200 mg | Period 3: Part B 50 mg | Period 3: Part B 100 mg | Period 3: Part B 200 mg | Period 4: Part C
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 57
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 38
Not completed — Study Terminated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 30
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Site Terminated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: The ITT Analysis Set included all randomized participants regardless of Treatment Period eligibility or completion. The ITT Analysis Set was the basis for demographics, baseline characteristics, and efficacy analyses.
Groups:
- Placebo: tablet
- Tildacerfont 50 mg: 50 mg
- Tildacerfont 100 mg: 100 mg
- Tildacerfont 200 mg: 200 mg
- Total: Total of all reporting groups
Arm/Group | Placebo | Tildacerfont 50 mg | Tildacerfont 100 mg | Tildacerfont 200 mg | Total
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (12.03) | 29.1 (11.55) | 31.5 (8.29) | 35.1 (11.36) | 32.3 (10.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 12 | 16 | 51
  Male | 12 | 13 | 12 | 8 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 3 | 4
  Not Hispanic or Latino | 23 | 24 | 24 | 21 | 92
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 1 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 21 | 22 | 22 | 19 | 84
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.46 (9.29) | 31.27 (7.675) | 30.98 (7.521) | 30.25 (4.453) | 30.99 (7.23)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 95.8 (17.074) | 98.78 (19.135) | 97.98 (19.148) | 99.31 (12.407) | 97.968 (16.941)
Daily dose of Glucocorticoid [Mean (Standard Deviation); unit: mg in hydrocortisone equivalent(s)] | 26.9 (7.59) | 29.1 (10.83) | 25.4 (6.71) | 26.7 (8.94) | 27.025 (8.518)
Glucocorticoid BSA Based Dose [Mean (Standard Deviation); unit: mg in hydrocortisone equivalent(s)/m^2] | 13.97 (4.198) | 14.62 (4.880) | 13.52 (4.117) | 14.21 (12.5) | 14.08 (6.424)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 118.3 (10.08) | 117.5 (9.54) | 115.0 (10.46) | 120.4 (13.71) | 117.8 (10.946)
Diastolic blood pressure [Median (Standard Deviation); unit: mmHg] | 78.1 (9.15) | 76.4 (7.03) | 77.6 (8.41) | 76.8 (10.27) | 77.225 (8.715)
HbA1c [Mean (Standard Deviation); unit: % of Hemoglobin] | 5.18 (0.215) | 5.14 (0.255) | 5.33 (0.944) | 5.27 (0.218) | 5.23 (0.408)
Fasting glucose [Mean (Standard Deviation); unit: mg/dL] | 89.1 (11.94) | 91.1 (9.57) | 91.4 (8.36) | 90.8 (10.03) | 90.6 (9.975)
Fasting insulin [Mean (Standard Deviation); unit: uIU/mL] | 10.32 (5.491) | 16.72 (9.896) | 15.77 (15.89) | 16.45 (11.004) | 14.815 (10.57)
Homeostatic model assessment of insulin resistance (HOMA-IR) [Mean (Standard Deviation); unit: units on a scale] — HOMA-IR stands for "Homeostatic Model Assessment for Insulin Resistance" and it is calculated from fasting glucose and fasting insulin. HOMA-IR = (Insulin (mU/L) × Glucose (mg/dL)) / 405. Less than 1 means you are insulin-sensitive (optimal), greater than 1.9 indicates early insulin resistance, and greater than 2.9 indicates significant insulin resistance.
  units on a scale | 2.33 (1.376) | 3.84 (2.507) | 3.66 (3.90) | 3.79 (2.774) | 3.405 (2.639)
Total cholesterol [Mean (Standard Deviation); unit: mg/dL] | 169.3 (41.62) | 158.6 (42.08) | 152.2 (29.15) | 179.3 (40.75) | 164.85 (38.4)
LDL [Mean (Standard Deviation); unit: mg/dL] | 91.2 (29.91) | 88.3 (32.22) | 85.8 (21.75) | 105.6 (31.67) | 92.725 (28.888)
HDL [Mean (Standard Deviation); unit: mg/dL] | 56.7 (18.85) | 44.0 (16.34) | 49.4 (11.14) | 49.3 (15.52) | 49.85 (15.463)
Triglycerides [Mean (Standard Deviation); unit: ng/dL] | 107.4 (52.48) | 131.3 (85.37) | 85.1 (33.35) | 133.0 (91.02) | 114.2 (65.555)
Cortisol [Mean (Standard Deviation); unit: ug/dL] | 2.63 (3.492) | 7.08 (9.382) | 1.29 (0.854) | 1.07 (1.071) | 3.018 (3.6998)
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 9 | 10 | 6 | 9 | 34
  Europe | 9 | 11 | 16 | 6 | 42
  Rest of World | 6 | 3 | 2 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Effect of Tildacerfont in Reducing A4 in Participants With Classic Congenital Adrenal Hyperplasia (CAH) Over 12 Weeks
Description: Assessment of dose response for change from baseline in log A4 after 12 weeks on double-blind placebo-controlled treatment (Week 18)
Time Frame: Baseline and 12 weeks of treatment (Week 18)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: log(ng/dL)
Arm/Group | Placebo | Tildacerfont 50 mg | Tildacerfont 100 mg | Tildacerfont 200 mg
Number analyzed (Participants) | 24 | 24 | 24 | 24
log(ng/dL) | 38.7 (307.38) | -49.0 (449.02) | 147.2 (661.2) | -10.4 (408.68)

2. Secondary Outcome: To Evaluate the Effect of Tildacerfont in Reducing A4 in Participants With Classic CAH Over 12 Weeks
Description: Absolute change from baseline in A4 as determined via application of the delta theorem to the log scale analysis results after 12 weeks on double-blind, placebo-controlled treatment (Week 18). Results show mean Treatment Effect of Dose vs Placebo. A negative value represents a reduction in absolute concentration compared to baseline.
Time Frame: 12 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Placebo | Tildacerfont 50 mg | Tildacerfont 100 mg | Tildacerfont 200 mg
Number analyzed (Participants) | 24 | 23 | 24 | 24
ng/dL | 0 (0) | -29.5 (106.26) | 39.1 (108.66) | -23.2 (107.72)

3. Secondary Outcome: To Evaluate the Effect of Tildacerfont in Reducing A4 in Participants With Classic CAH Over 12 Weeks
Description: Change from baseline in A4 as assessed on the log scale after 12 weeks on double-blind, placebo-controlled treatment (Week 18). Results show mean % of Treatment Effect of Dose vs Placebo. A negative value represents a % reduction from baseline.
Time Frame: 12 weeks
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Placebo | Tildacerfont 50 mg | Tildacerfont 100 mg | Tildacerfont 200 mg
Number analyzed (Participants) | 24 | 23 | 24 | 24
percentage | 0 [0 to 0] | -3.3 [-23.7 to 22.7] | 4.3 [-17.4 to 31.8] | -2.6 [-23.3 to 23.9]

4. Secondary Outcome: To Evaluate the Effect of Tildacerfont in Reducing 17-OHP in Participants With Classic CAH Over 12 Weeks
Description: Change from baseline in 17-OHP as assessed on the log scale after 12 weeks on double-blind, placebo-controlled treatment (Week 18). A negative value represents a % reduction from baseline.
Time Frame: 12 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Tildacerfont 50 mg | Tildacerfont 100 mg | Tildacerfont 200 mg
Number analyzed (Participants) | 24 | 20 | 22 | 20
percent change | 215.6 (6165.61) | 644.2 (6580.01) | 3564.6 (7490.8) | -753.7 (5698.97)
Statistical Analysis 1: Comparison: Tildacerfont 50 mg vs Tildacerfont 100 mg vs Tildacerfont 200 mg; Test type: Other — Assessment of dose response for change from baseline in log 17-OHP after 12 weeks on double-blind, placebo-controlled treatment (Week 18). Results were obtained by using a repeated measures random coefficient mixed-effects model and are reported as the -2loglikelihood results for both the full (including interaction terms) and reduced (excluding interaction terms) models; p = 0.8051, Mixed Models Analysis — Dose response p-value; The result for the -2loglikelihood full model was -580.2550766 log(ng/dL) and -583.2846546 log(ng/dL) for the reduced model

5. Secondary Outcome: To Evaluate the Effect of Tildacerfont in Reducing 17-OHP in Participants With Classic CAH Over 12 Weeks
Description: Absolute change from baseline in 17-OHP as determined via application of the delta theorem to the log scale analysis results after 12 weeks on double-blind, placebo-controlled treatment (Week 18). Results show mean Treatment Effect of Dose vs Placebo. A negative value represents a reduction in absolute concentration compared to baseline.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Placebo | Tildacerfont 50 mg | Tildacerfont 100 mg | Tildacerfont 200 mg
Number analyzed (Participants) | 24 | 23 | 24 | 24
ng/dL | 0 (0) | 355.9 (2179.63) | 22.6 (2120.47) | -250.8 (2153.59)

ADVERSE EVENTS:
Time Frame: 60 weeks (12 weeks Part A, 12 weeks Part B, 46 weeks Part C)
Groups:
- Period 2: Part A 50 mg; Period 3: Part B 50 mg: tildacerfont tablet administered daily via oral tablet for 12 weeks at 50 mg
- Period 2: Part A 100 mg; Period 3: Part B 100 mg: tildacerfont tablet administered daily via oral tablet for 12 weeks at 100 mg
- Period 2: Part A 200 mg: tildacerfont tablet administered daily via oral tablet for 12 weeks at 200 mg
- Period 3: Part B 200 mg: Tildacerfont tablet administered daily via oral tablet for 12 weeks 200 mg
Arm/Group | Period 1: Placebo | Period 2: Part A 50 mg | Period 2: Part A 100 mg | Period 2: Part A 200 mg | Period 3: Part B 50 mg | Period 3: Part B 100 mg | Period 3: Part B 200 mg | Period 4: Part C
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/1 | 0/44 | 0/41 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/24 | 1/24 | 0/24 | 0/1 | 2/44 | 0/41 | 1/57
Other Adverse Events (participants affected / at risk) | 17/24 | 16/24 | 20/24 | 16/24 | 0/1 | 26/44 | 17/41 | 38/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Placebo (N=24) | Period 2: Part A 50 mg (N=24) | Period 2: Part A 100 mg (N=24) | Period 2: Part A 200 mg (N=24) | Period 3: Part B 50 mg (N=1) | Period 3: Part B 100 mg (N=44) | Period 3: Part B 200 mg (N=41) | Period 4: Part C (N=57)
COVID-19 (Infections and infestations) | NA | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (Nervous system disorders) | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0)
Status Epilepticus (Nervous system disorders) | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal Pneumonia (Infections and infestations) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal septum deviation (Musculoskeletal and connective tissue disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Placebo (N=24) | Period 2: Part A 50 mg (N=24) | Period 2: Part A 100 mg (N=24) | Period 2: Part A 200 mg (N=24) | Period 3: Part B 50 mg (N=1) | Period 3: Part B 100 mg (N=44) | Period 3: Part B 200 mg (N=41) | Period 4: Part C (N=57)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 6 (6)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 10 (10)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 5 (5)
Asthenia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Influenza like illness (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland mucocoele (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 4 (4) | 5 (5) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Status epipticus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Asymptomatic COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Temperature regulation disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trigger fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Emotional distress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fear of Injection (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Social communication disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressive symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foreign body in throat (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood prolactin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood follicle stimulating hormone decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood luteinising hormone decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Total bile acids increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insulin resistance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food Intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased apetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tetany (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oligomenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polymenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal mass (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thyroiditis subacute (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye Swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Family stress (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT04457336/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/36/NCT04457336/SAP_001.pdf